CLINICAL TRIAL: NCT00562393
Title: Effects of Excess Energy Intake on Metabolic Risk
Acronym: EXCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Garvan Institute of Medical Research (Other)
Responsible Party: Principal Investigator, Dr Jerry Greenfield, Head of Endocrinology Department St Vincent's Hospital Sydney, Garvan Institute of Medical Research
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: EXCESS; 427639
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Overfeeding (Experimental): 4 weeks of 1250 kcal added daily
  Interventions: Other: Nutritional

INTERVENTIONS:
Other: Nutritional — Overfeeding high fat diet for 28 days

SUMMARY:
The prevalence of obesity has reached epidemic proportions and is associated with the development of insulin resistance and type 2 diabetes (T2DM). A unifying theme has emerged over the past few years suggesting that lipid oversupply to metabolic organs responsible for glucose regulation leads to insulin resistance. Fitting with this, we and others have shown that increased lipid accumulation within skeletal muscle and/or liver is associated with impaired glucose uptake. However, the underlying mechanisms that mediate changes in muscle lipid metabolism are not yet known. The overall aim of this project is to examine metabolic effects of experimental weight gain in lean and overweight individuals with and without a genetic predisposition to type 2 diabetes. We hypothesise that lean subjects will increase fatty acid oxidation and upregulate mitochondrial oxidative capacity in muscle following overfeeding to protect against body weight gain and insulin resistance, but overweight subjects with a genetic predisposition to T2DM will have a defect in this ability.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (<60 min formal exercise per week)
* Aged 20-65 years

Exclusion Criteria:

* Personal history of diabetes, cardiovascular disease or hypertension
* Recent weight change (larger than 4kg in the past 3 months)
* Smoking
* Regular use of medications, except oral contraceptives
* Individuals with alcoholism or other substance abuse
* Pregnancy or lactation, women who are planning to become pregnant or who are not using adequate measures of birth control.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Insulin sensitiviy by hyperinsulinemic clamp | 28-days

SECONDARY OUTCOMES:
Fat oxidation (whole body RQ and C-14 palmitate), mitochondrial function | 28-days

CONTACTS AND LOCATIONS:
Overall Officials: Leonie K Heilbronn, PhD, Principal Investigator — Garvan Institute; Lesley M Campbell, MBBS, Principal Investigator — Garvan Insititute
Locations (1):
- Garvan Institute of Medical Research, Darlinghurst, New South Wales, Australia

REFERENCES:
- [Result] Tam CS, Viardot A, Clement K, Tordjman J, Tonks K, Greenfield JR, Campbell LV, Samocha-Bonet D, Heilbronn LK. Short-term overfeeding may induce peripheral insulin resistance without altering subcutaneous adipose tissue macrophages in humans. Diabetes. 2010 Sep;59(9):2164-70. doi: 10.2337/db10-0162. Epub 2010 Jun 14. PMID 20547978
- [Result] Samocha-Bonet D, Campbell LV, Viardot A, Freund J, Tam CS, Greenfield JR, Heilbronn LK. A family history of type 2 diabetes increases risk factors associated with overfeeding. Diabetologia. 2010 Aug;53(8):1700-8. doi: 10.1007/s00125-010-1768-y. Epub 2010 May 12. PMID 20461357
- [Result] Sato K, Samocha-Bonet D, Handelsman DJ, Fujita S, Wittert GA, Heilbronn LK. Serum sex steroids and steroidogenesis-related enzyme expression in skeletal muscle during experimental weight gain in men. Diabetes Metab. 2014 Dec;40(6):439-44. doi: 10.1016/j.diabet.2014.03.006. Epub 2014 Apr 30. PMID 24792219
- [Result] Samocha-Bonet D, Tam CS, Campbell LV, Heilbronn LK. Raised circulating fetuin-a after 28-day overfeeding in healthy humans. Diabetes Care. 2014;37(1):e15-6. doi: 10.2337/dc13-1728. No abstract available. PMID 24356603
- [Result] Heilbronn LK, Coster AC, Campbell LV, Greenfield JR, Lange K, Christopher MJ, Meikle PJ, Samocha-Bonet D. The effect of short-term overfeeding on serum lipids in healthy humans. Obesity (Silver Spring). 2013 Dec;21(12):E649-59. doi: 10.1002/oby.20508. Epub 2013 Jul 29. PMID 23640727
- [Result] Heilbronn LK, Campbell LV, Xu A, Samocha-Bonet D. Metabolically protective cytokines adiponectin and fibroblast growth factor-21 are increased by acute overfeeding in healthy humans. PLoS One. 2013 Oct 18;8(10):e78864. doi: 10.1371/journal.pone.0078864. eCollection 2013. PMID 24205333
- [Result] Samocha-Bonet D, Campbell LV, Mori TA, Croft KD, Greenfield JR, Turner N, Heilbronn LK. Overfeeding reduces insulin sensitivity and increases oxidative stress, without altering markers of mitochondrial content and function in humans. PLoS One. 2012;7(5):e36320. doi: 10.1371/journal.pone.0036320. Epub 2012 May 7. PMID 22586466
- [Derived] Elshorbagy AK, Samocha-Bonet D, Jerneren F, Turner C, Refsum H, Heilbronn LK. Food Overconsumption in Healthy Adults Triggers Early and Sustained Increases in Serum Branched-Chain Amino Acids and Changes in Cysteine Linked to Fat Gain. J Nutr. 2018 Jul 1;148(7):1073-1080. doi: 10.1093/jn/nxy062. PMID 29901727